CLINICAL TRIAL: NCT03822689
Title: The Influences of Different Type of Ventilation Breathing Tube Among Children and Neonate Under General Anesthesia
Brief Title: Comparison of Ventilation Tubes Among Anesthetized Pediatrics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Institutional Review Board did not approve
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Chung,Huang, attending physician, department of anesthesiology, Mackay Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19MMHIS025e
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Ventilation
Keywords: pediatric; Ventilation breathing tube; End-Tidal Carbon Dioxide; Heart rate; tidal volume; blood temperature

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gas flow:2L (Active Comparator): use different type ventilator breathing tube as follow Ventilator breathing tube F2220-M: Folding; D: 22mm; L:2.0M Ventilator breathing tube F2216-M: Folding; D: 22mm; L:1.6M Ventilator breathing tube F1520-M: Folding; D: 15mm; L:2.0M Ventilator breathing tube F1516-M: Folding; D: 15mm; L:1.6M Ventilator breathing tube U1016-M: Unfolding; D: 10mm; L:1.6M Ventilator breathing tube U1516-M: Unfolding; D: 15mm; L:1.6M Ventilator breathing tube CA20-.M: Co-axis; L:2.0M Ventilator breathing tube CA16- M: Co-axis; L:1.6M
  Interventions: Device: Ventilator breathing tube F2220; Device: Ventilator breathing tube F2216; Device: Ventilator breathing tube F1520; Device: Ventilator breathing tube F1516; Device: Ventilator breathing tube U1016; Device: Ventilator breathing tube U1516; Device: Ventilator breathing tube CA20; Device: Ventilator breathing tube CA16
- Gas flow:5L (Active Comparator): use different type ventilator breathing tube as follow Ventilator breathing tube F2220-M: Folding; D: 22mm; L:2.0M Ventilator breathing tube F2216-M: Folding; D: 22mm; L:1.6M Ventilator breathing tube F1520-M: Folding; D: 15mm; L:2.0M Ventilator breathing tube F1516-M: Folding; D: 15mm; L:1.6M Ventilator breathing tube U1016-M: Unfolding; D: 10mm; L:1.6M Ventilator breathing tube U1516-M: Unfolding; D: 15mm; L:1.6M Ventilator breathing tube CA20-.M: Co-axis; L:2.0M Ventilator breathing tube CA16- M: Co-axis; L:1.6M
  Interventions: Device: Ventilator breathing tube F2220; Device: Ventilator breathing tube F2216; Device: Ventilator breathing tube F1520; Device: Ventilator breathing tube F1516; Device: Ventilator breathing tube U1016; Device: Ventilator breathing tube U1516; Device: Ventilator breathing tube CA20; Device: Ventilator breathing tube CA16

INTERVENTIONS:
Device: Ventilator breathing tube F2220 — M: Folding D: 22mm; L: 2.0M
Device: Ventilator breathing tube F2216 — M: Folding; D: 22mm; L:1.6M
Device: Ventilator breathing tube F1520 — M: Folding; D: 15mm; L:2.0M
Device: Ventilator breathing tube F1516 — M: Folding; D: 15mm; L:1.6M
Device: Ventilator breathing tube U1016 — M: Unfolding; D: 10mm; L:1.6M
Device: Ventilator breathing tube U1516 — M: Unfolding; D: 15mm; L:1.6M
Device: Ventilator breathing tube CA20 — M: Co-axis; L:2.0M
Device: Ventilator breathing tube CA16 — M: Co-axis; L:1.6M

SUMMARY:
To discover whether different types of ventilation breathing tube influence ventilation effect of children/ neonate, the investigators analysis tidal volume, end tidal carbon dioxide, compliance among children and neonate under general anesthesia. The study compares eight ventilator breathing tube of different length, diameter, material of the ventilator breathing tube. Besides, the investigators also make an approach verify the change of body temperate under different gas flow(2L, and 5L).

DETAILED DESCRIPTION:
In previous research, initial mechanical ventilator settings about children were as following: 1.tidal volume 6 to 10 ml/kg of ideal body weight; 2.delta pressures of respiratory pressure should be <10 cmH2O in healthy patients; 3. respiratory pressures could be kept less than 28 to 30 cmH2O in patient with lung injury; 4. positive end-expiratory pressure was necessary, although the optimal level is unknown.

However, few researches discussed about Influences of different types of ventilation breathing tube. The investigators want to clarify the character about length, diameter, and material of the ventilation breathing tube under the ventilation system in relation to tidal volume, end tidal carbon dioxide, compliance among children and neonate.

During this study, the participants will be 100 children who were ASA class1, 2 and performed non-emergency, non-cardiac surgery, who will receive general anesthesia . The participants will divide into three groups according to different body weights (Group N: <4.5kg; Group T: 4.5~20kg; Group C: >20kg), and would receipt total eight type of ventilator breathing tube test. Primary outcome will be the difference of tidal volume, end tidal carbon dioxide and compliance. Besides, secondary outcome will be the change of body temperate under different gas flow (2L, and 5L).

ELIGIBILITY:
Inclusion Criteria:

* with American Society of Anesthesiologists (ASA) physical status classification 1&2
* undergo elective surgery
* intubation

Exclusion Criteria:

* Cardiac-pulmonary surgery
* Had respiratory related disease

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Tidal volume | From: 1 minute after endotracheal intubation, and vital signs include heart rate, blood pressure, EtCO2 did not change over 30%. To: eight types of tubes have already tested, up to 30 minutes after beginning
  compared tidal volume besides different ventilation breathing tube
End tidal carbon dioxide | From: 1 minute after endotracheal intubation, and vital signs include heart rate, blood pressure, EtCO2 did not change over 30%. To: eight types of tubes have already tested, up to 30 minutes after beginning
  compared End tidal carbon dioxide besides different ventilation breathing tube

SECONDARY OUTCOMES:
Body temperate | From: 1 minute after endotracheal intubation, and vital signs include heart rate, blood pressure, EtCO2 did not change over 30%. To: eight types of tubes have already tested, up to 30 minutes after beginning
  compared Body temperate about different gas flow(2L,5L)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chung Huang, MD, Study Director — Mackay Memorial Hospital
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman JM. Optimal ventilation of the anesthetized pediatric patient. Anesth Analg. 2015 Jan;120(1):165-175. doi: 10.1213/ANE.0000000000000472. PMID 25625261
- [Background] Kneyber MC. Intraoperative mechanical ventilation for the pediatric patient. Best Pract Res Clin Anaesthesiol. 2015 Sep;29(3):371-9. doi: 10.1016/j.bpa.2015.10.001. Epub 2015 Oct 14. PMID 26643101
- [Background] Glenski TA, Diehl C, Clopton RG, Friesen RH. Breathing circuit compliance and accuracy of displayed tidal volume during pressure-controlled ventilation of infants: A quality improvement project. Paediatr Anaesth. 2017 Sep;27(9):935-941. doi: 10.1111/pan.13164. Epub 2017 May 15. PMID 28504341
- [Background] von Goedecke A, Brimacombe J, Hormann C, Jeske H-, Kleinsasser A, Keller C. Pressure support ventilation versus continuous positive airway pressure ventilation with the ProSeal laryngeal mask airway: a randomized crossover study of anesthetized pediatric patients. Anesth Analg. 2005 Feb;100(2):357-360. doi: 10.1213/01.ANE.0000143563.39519.FD. PMID 15673856